CLINICAL TRIAL: NCT01572766
Title: Impact of the FRAX Assessment on Physician and Patient Treatment Behavior
Brief Title: Effect of Assessing Risk for Osteoporosis on Physician and Patient Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: Warner Chilcott (Industry)
Responsible Party: Principal Investigator, Hildegarde J. Berdine, Associate Professor of Pharmacy Practice, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Osteo Prevention
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteoporosis; Pharmacist; Behavior Change; FRAX; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FRAX Assessment (Active Comparator): FRAX Assessment Tool administered by a pharmacist. This group also receives a heel ultrasound and pharmacist counseling.
  Interventions: Other: FRAX Assessment Tool
- Control group (No Intervention): Control group receives heel ultrasound and pharmacist counseling

INTERVENTIONS:
Other: FRAX Assessment Tool — FRAX Assessment Tool is designed to assess risk for fracture based on country of origin, race, and other factors.
  Other Names: WHO FRAX Risk Assessment Tool
  Arms: FRAX Assessment

SUMMARY:
The study seeks to determine the impact of assessing risk for osteoporosis in women on patient and physician behaviors through a pharmacist directed osteoporosis screening program. Women will be offered a heel ultrasound to screen for their bone density and may or may not be asked questions about their risk for bone fracture. Pharmacists will counsel and educate all women on ways to prevent the onset of osteoporosis. Women will be telephoned three months after the screening and asked a series of 10 questions to follow up on decisions made by their physicians or changes made to their health behaviors related to bone health.

DETAILED DESCRIPTION:
A maximum of 90 participants will be recruited and randomized to the FRAX® assessment intervention group or the control group to a total of 45 participants in each group. The number of participants was chosen based on the simple randomized design of the study and use of basic statistics (versus regression analysis). Subjects will be recruited from the employee population of Duquesne University, clients visiting the Spirit of Health mobile health unit, and the downtown Pittsburgh community and surrounding neighborhoods of Duquesne University. Participants will be recruited through posted flyers at these various screening venues. Data collected will be the T-score at baseline screening in both groups. The percent risk for fracture as determined by the FRAX® tool will be determined for the intervention group. After 3 months have elapsed, a questionnaire will be administered via telephone to both the intervention and control groups, a series of 12 yes/no questions. Fisher's exact test will be used to analyze the data. Data collected will be nominal data with n in each group at 45 for a total of 90 participants. Descriptive statistics will also be employed.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

1. Postmenopausal female participants over the age of 45 years up to and including 65 years of age. The participant will be required to have a medical doctor and covered by an insurance plan in case a DXA-scan is ordered by the physician.
2. Ability to be screened at the Center for Pharmacy Care or at other community screenings on the Achilles® heel ultrasound bone densitometer.
3. After heel ultrasound is conducted, include those individuals as participants in the study who present with a T-score equal to or less than -1.0.

Exclusion Criteria:

1. Unable to participate in the follow-up survey conducted over the telephone.
2. Age less than 45 years or over 65 years.
3. Any individual currently taking biphosphonates for osteoporosis treatment.
4. After heel ultrasound is conducted, if T-score is greater than -1.0.
5. Males

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Behavior Change | After 3 months or greater from screening.
  Patient Health behavior changes included beginning exercise, initiating calcium and vitamin D supplements, talking with physician about osteoporosis prevention, screening by DXA scan, changing dietary intake of calcium; physician behavior changes included ordering a DXA scan, ordering vitamin D blood levels, initiating drug treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hildegarde J Berdine, PharmD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University Center for Pharmacy Care, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Watts NB. The Fracture Risk Assessment Tool (FRAX(R)): applications in clinical practice. J Womens Health (Larchmt). 2011 Apr;20(4):525-31. doi: 10.1089/jwh.2010.2294. Epub 2011 Mar 25. PMID 21438699
- [Background] Elias MN, Burden AM, Cadarette SM. The impact of pharmacist interventions on osteoporosis management: a systematic review. Osteoporos Int. 2011 Oct;22(10):2587-96. doi: 10.1007/s00198-011-1661-7. Epub 2011 Jul 1. PMID 21720894
- [Result] Izuora KE, Alazraki N, Byrd-Sellers J, Tangpricha V, Nanes MS. Fracture assessment tool risk scores in bone density reports do not change physician prescribing behavior for osteoporosis. Am J Med Sci. 2011 Jul;342(1):5-8. doi: 10.1097/MAJ.0b013e31820aba02. PMID 21412137
- See also: National Osteoporosis Foundation — http://www.nof.org
- See also: World Health Organization Fracture Risk Assessment Tool — http://www.shef.ac.uk/FRAX